CLINICAL TRIAL: NCT02255149
Title: Vertical Ridge Augmentation Using Titanium Mesh and Allograft in Posterior Mandible: A Feasibility Study
Brief Title: A Feasibility Study for Growth Bone Vertically With Titanium Mesh and Allograft in Lower Posterior Jaw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00053796
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone/Mesh (Experimental): Allograft and Titanium mesh will be used to grow jaw bone vertically.
  Interventions: Device: Bone/Mesh

INTERVENTIONS:
Device: Bone/Mesh — A titanium mesh (Ti-Mesh) that is more porous than other materials will be placed in order to hold a spot for the bone particles to grow.

SUMMARY:
This study will involve placing donor bone into the back of lower jaw then covering with a newly designed titanium mesh. The mesh will then stay in the mouth for 4 months before it will be removed. Implants will be placed in the newly formed bone.

The goal of this study is to test how well using a newly designed titanium mesh and bone particles can grow bone in the back of the lower jaw. The investigators are also checking if the newly formed bone will stay around implants that will have been in use for 12 months.

DETAILED DESCRIPTION:
Inclusion Criteria

* Patients are at least 18 years old
* At least two adjacent back teeth in the lower jaw are missing
* No medical contraindication to dental surgery
* Inadequate vertical ridge height at edentulous region (less than 10mm)

Exclusion Criteria

* Unstable systemic diseases or conditions that would compromise the healing potential
* Patients with osseous metabolic disorders (e.g., osteoporosis, Paget's disease etc.)
* Patients who are pregnant or expect to get pregnant
* Patients with unstable dental disease (e.g. caries and periodontitis) in the surgical sextant

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients (ASA I or II)
* Non-smoker or light smokers (< 10 cigarettes per day)
* Good oral health (FMPS and FMBS <20%)
* At least two adjacent mandibular posterior teeth are missing
* Inadequate vertical ridge height at edentulous region (less than 10mm)
* Missing teeth for ≥ 3 months

Exclusion Criteria:

* Unstable and complicated systemic diseases or chronic disorders precluding surgical procedures
* Systemic diseases with compromised healing potentials (Uncontrolled Diabetes Mellitus, HIV infections, etc.)
* Bone disorders (Hyperparathyroidism, Osteoporosis, Paget's Disease)
* Pregnant or expecting to become pregnant
* Currently smoking (≥ 10 cigarettes/day)
* Poor oral hygiene (≥20% Modified O'Leary Plaque Index)
* Severe grinding, clenching, TMJ disorder
* Untreated dental disease (periodontitis, caries, abscesses) in the research quadrant
* Teeth exhibiting periapical pathology or purulence (symptomatic) in the research quadrant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsun-Liang Chan, DDS, MS, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan HL, Benavides E, Tsai CY, Wang HL. A Titanium Mesh and Particulate Allograft for Vertical Ridge Augmentation in the Posterior Mandible: A Pilot Study. Int J Periodontics Restorative Dent. 2015 Jul-Aug;35(4):515-22. doi: 10.11607/prd.1980. PMID 26133141

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone/Mesh
Started | 10
Completed | 5
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by PI | 1
Not completed — Implant Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bone/Mesh
Number analyzed (Participants) | 10
Age, Customized [Number; unit: years]
  >=18 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Bone height [Mean (Full Range); unit: millimeters] | 9.8 [7.2 to 12.9]

OUTCOME MEASURES:

1. Primary Outcome: Bone Height
Description: Diameter of the bone measured from the alveolar crest to the inferior alveolar nerve after the grafting procedures from CBCT images.
Time Frame: 5 months
Measure: Mean (Full Range); unit: millimeters
Arm/Group | Bone/Mesh
Number analyzed (Participants) | 5
millimeters | 12.2 [8.0 to 14.4]

ADVERSE EVENTS:
Time Frame: 2 years 6 months
Arm/Group | Bone/Mesh
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone/Mesh (N=10)
Implant Failure (Surgical and medical procedures) | 2 (3)
Mesh Exposure/Removal (Surgical and medical procedures) | 6 (6)
Headache (General disorders) | 1 (1)
Hypoxic Tissue (Blood and lymphatic system disorders) | 1 (1)
Lack of Bone Growth (Surgical and medical procedures) | 1 (1)
Wound Opening at Mesh site (Surgical and medical procedures) | 2 (2)
Soft Tissue Dehiscence (Surgical and medical procedures) | 1 (1)
Soreness on Tongue (General disorders) | 1 (1)
Throbbing Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No